CLINICAL TRIAL: NCT02773420
Title: HET Bipolar System: Validation of a New Minimally Invasive Outpatient Treatment for Symptomatic Hemorrhoids
Brief Title: HET Bipolar System: Validation of Outpatient Hemorrhoid Treatment
Acronym: HET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Johan Nordenstam, Assistant Professor of Surgery, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0701; ISR-2015-10644 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HET application arm (Experimental): Patients with grade I-II internal hemorrhoids will undergo HET application
  Interventions: Procedure: HET Application

INTERVENTIONS:
Procedure: HET Application — The HET device is a modified anoscope equipped with LED lighting, a tissue clamping mechanism and a bipolar energy source used to treat multiple hemorrhoidal columns in one sitting. Three columns of hemorrhoids were treated with 2 heat energy applications per column

SUMMARY:
Purpose: The current study aims to evaluate the safety and effectiveness of the HET™ Bipolar System (Medtronic, Boulder, CO) for the treatment of grade I-II hemorrhoids in a prospective pilot study. This device was evaluated retrospectively in a limited cohort of 23 patients previously.

Methods: Patients seen at a colorectal clinic in a single institution with grade I-II hemorrhoids are offered to participate in a prospective pilot trial. The HET device is a modified anoscope equipped with LED lighting, a tissue clamping mechanism and a bipolar energy source used to treat multiple hemorrhoidal columns in one sitting. Three columns of hemorrhoids are treated with 2 heat energy applications per column. The primary outcome is the treatment effect on hemorrhoid symptoms of bleeding, pain, prolapse, itching, and soiling. This is measured with a patient completed questionnaire documenting each symptom's frequency from 0 to 3 (i.e. 0 is < 1x/month; 3 is daily) before therapy and at 3 weeks and 6 month follow-up. Post-treatment pain scores were recorded using the visual analog scale (VAS).

DETAILED DESCRIPTION:
HET Bipolar System: Validation of Outpatient Hemorrhoid Treatment

Introduction: This study will evaluate the effectiveness of treatment of Grade I-II hemorrhoids with the novel HET Bipolar System (Medtronic, Boulder, Co.). This device is a modified anoscope equipped with LED lighting, tissue clamping mechanism and bipolar energy device. It is inserted in the anus under direct vision targeting the tissue proximal to the hemorrhoid, which is placed within the treatment window and clamped. The bipolar energy device is activated to ligate the feeding hemorrhoidal vessels, essentially disrupting the blood supply to the hemorrhoid. The only published evaluation of this device to date is a retrospective analysis of the safety and efficacy of the device in 23 patients (1).

There is no prospective study of this device and its effectiveness in the literature. The investigators aim to evaluate the efficacy of this device, defined as decrease in symptoms and/or recurrence, of Grade I-II hemorrhoids through a prospective study consisting of 30 patients. Other non invasive means of treating hemorrhoids range from sclerotherapy to rubber band ligation, which often requires multiple treatments and can cause some discomfort. The investigators aim to study HET Bipolar treatment of hemorrhoids to offer another validated minimally invasive option for the treatment of symptomatic hemorrhoids in the outpatient setting.

Research Design and Method: The investigators will enroll a total of 30 subjects. Participating patients,18 years of age and older, will be undergoing treatment with the HET bipolar system for symptomatic Grade I and II hemorrhoids. Please note that the HET bipolar system is used as part of standard of care and participants will receive the treatment regardless of this research. The subjects will be identified and recruited by University of Illinois at Chicago Department of Colorectal Surgery faculty via clinic appointments in the Outpatient Care Center, 1801 W. Taylor St, Suite 3F, Chicago, Il 60612. Informed consent will be provided at the clinic in regards to participation in the study. Refusal to participate will not influence treatment options presented or deemed necessary for the subject's condition. A pretreatment hemorrhoid symptom questionnaire will be completed by each patient. In developing our questionnaire the investigators examined the only validated hemorrhoidal symptom questionnaire in the literature, the Sodergren Score (2) and also various others (3). The Sodergren score offers a theoretical basis, however the investigators chose to develop a questionnaire secondary to the need for inclusion of bleeding symptoms of hemorrhoids. While subjects are undergoing treatment, the investigators will record timing of treatment, number of hemorrhoids treated, and energy application timing. Immediately after the treatment, the patients will describe how painful the procedure was using the Visual Analog Scale (VAS). The questionnaire will take 5-10 minutes to complete. Patients will be seen for follow up outpatient clinic visits at 2-3 weeks and at 8-12 weeks post procedure. At follow up, the patients will be given a post-treatment questionnaire regarding symptoms of hemorrhoids (this is the same questionnaire as the pre-treatment questionnaire). The questionnaire assigns each of the five cardinal symptoms of hemorrhoids with a number from 0 to 3 with 3 being the most severe symptom. After tallying the five symptom scores, a total from 0 (no symptoms) to 15 (severe symptoms) will be assigned to each patient's overall symptoms. In addition, patients will be given a journal to record their daily pain for 14 consecutive days, day 21 and day 56 using the Visual Analog Scale (VAS). This is to more accurately record pain, as the questionnaire does not include a VAS score component. Patients who are unable to come for follow up visits will be interviewed over the phone by one of the investigators and the relevant data, i.e. the questionnaire and pain score, will be obtained during this phone conversation. For patients following up over the phone, a phone script will be created in addition to the questionnaire. The total number of visits/encounters is 3 and will take place during regular clinic visit appointments. The difference between pre treatment and post treatment scores will be representative of the treatment effect.

Statistical Section:

Descriptive statistics will be used to describing the distribution of data. The Wilcoxon signed rank test will be used to examine the pre- and post- treatment symptom score difference. Paired two-sample t-test and McNemar's test will also be used to examine the pre- and post-treatment difference for other variables of interests.

Sample size justification:

Since the Wilcoxon signed rank test will be used to test the significant difference between pre- and post- treatment scores, the power calculation is based on the Wilcoxon signed rank test. At 80% power level, assuming correlation 0.2 between pre- and post- treatment scores, the sample size of 18 ensure minimum detectable difference in symptom score between pre- and post-treatment scores of 3. Thus, our sample size of 30 is appropriate.

Example: At 80% power level, assuming correlation 0.2 between pre- and post- treatment scores, the sample size of 18 ensure minimum detectable difference in symptom score between pre- and post-treatment scores of 3.

Expected Results/Conclusions: The investigators anticipate a significant decrease of hemorrhoidal symptoms, defined in this study as pain, pruritis, prolapse, soiling, and bleeding with the HET bipolar system, providing a validated outpatient minimally invasive treatment option for symptomatic hemorrhoids.

Benefits/Risks: There is no direct benefit to the subjects of this study. The main risk of this research is loss of confidentiality of information. The patient may experience mild anxiety or discomfort in providing information about their health and well-being. Records will be stored in an electronic data file on a password protected computer in a locked office. Master key will be kept in a separate file accessible only by the primary investigator.

Informed Consent:

Informed consent will be provided at the clinic in regards to participation in the study. Refusal to participate will not influence treatment options presented or deemed necessary for the subject's condition. Consent will be obtained by the primary investigator and/or research fellows who have experience and training in the explanation of the procedure, potential risks and benefits. The informed consent document will be stored in the subject's electronic medical record. If non-English speaking subjects are encountered, the informed consent will be translated by interpretation in the language of the subject.

Data and Safety Monitoring Plan:

This study poses minimal risk, the main risk being mild anxiety or loss of confidentiality of information. If problems arise they will be handled according to Institutional Review Board protocol.

Data Collection and Management Procedures:

Data procurement will be done electronically and incorporated in password protected encrypted server in a locked office. The master key will be kept in a separate file accessible only by the primary investigator.

Reporting Unanticipated Problems:

If any unanticipated problems arise they will be reported to University of Illinois at Chicago's Insitutional Review Board per defined protocol.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older.
2. Patients undergoing treatment for symptomatic hemorrhoids using the HET device

Exclusion Criteria:

1. All patients not included in Inclusion Criteria
2. Patients with inflammatory bowel disease, malignancy, anal fissures and those who are subject to anti-coagulation therapy with any drug other than aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
HET Treatment effect on hemorrhoid symptoms | 3 weeks to 6 months to 1 year
  The effect of HET on symptoms of bleeding, pain, prolapse, itching, and soiling.

SECONDARY OUTCOMES:
Pain associated with HET | Immediately to 3 weeks to 2 months
  Evaluation of pain associated with the procedure itself using visual analog scale for pain to record outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nordenstam, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Kantsevoy SV, Bitner M. Nonsurgical treatment of actively bleeding internal hemorrhoids with a novel endoscopic device (with video). Gastrointest Endosc. 2013 Oct;78(4):649-53. doi: 10.1016/j.gie.2013.05.014. Epub 2013 Jul 25. PMID 23891414
- [Result] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811
- [Result] Gerjy R, Lindhoff-Larson A, Sjodahl R, Nystrom PO. Randomized clinical trial of stapled haemorrhoidopexy performed under local perianal block versus general anaesthesia. Br J Surg. 2008 Nov;95(11):1344-51. doi: 10.1002/bjs.6379. PMID 18844245